CLINICAL TRIAL: NCT02321085
Title: The Comparison With Clinical Impacts on Functional Capacity and Symptom Improvement According to the Rhythm Control in Patients With Heart Failure and Recent Onset Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0811
Record Dates: First submitted 2014-11-20; First posted 2014-12-22 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure; Recent Onset Atrial Fibrillation
MeSH Terms: conditions — Heart Failure | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sinus Rhythm Control group (Active Comparator): 1. Start AAD right after evaluating for LA size, EF, LA thrombus, and presence of CAD during anticoagulation
  2. Cardioversion after 1 month
  3. Rhythm FU schedule (2012 ACC/AHA/ESC guidelines)
  4. If AF recur, RFCA
  Interventions: Procedure: Sinus Rhythm control
- Pulse Rate Control Group (Active Comparator): 1. No AAD, just anticoagulation
  2. HR control between 60~110bpm (with beta blocker, calcium channel blocker, digoxin)
  3. Without the treatment about antiarrhythmia and rhythm control, diffraction of rate control, the subject will be drop out for study.
  Interventions: Procedure: Pulse Rate control

INTERVENTIONS:
Procedure: Sinus Rhythm control
  Arms: Sinus Rhythm Control group
Procedure: Pulse Rate control
  Arms: Pulse Rate Control Group

SUMMARY:
Prospective randomized (rhythm control or rate control in heart failure patients with new onset atrial fibrillation) Objective of study 1. To analyze long term outcome of patients with heart failure with new onset atrial fibrillation according to the rhythm control 2. To analyze remodeling of atrium and ventricle by the new onset AF in heart failure patients 3. To analyze the change of LV function and functional capacity according to the rhythm in patients with HF and new onset AF

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Heart failure and Atrial fibrillation within 1year (20~80 years old)
2. LA diameter < 5mm
3. LVEF 20~49%
4. patients possible to anticoagulation and anti arrhythmic drug
5. Expected survival >1yr

Exclusion Criteria:

1. Impossible to anticoagulation or anti arrhythmic drug
2. valvular atrial fibrillation ( Mitral valve stenosis, Mitral valve plasty, valve replacement)
3. LV ejection fraction < 20%
4. Structural cardiac disease
5. Catheter ablation history for AF, maze surgery
6. patient with severe medical disease
7. Impossible to anticoagulation or anti arrhythmic drug

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
improvement of left ventricular function according to the rhythm control in patient with heart failure and new onset atrial fibrillation | 1 year
  ejection fraction change (echocardiography)
functional capacity according to the rhythm control in patient with heart failure and new onset atrial fibrillation | 1 year
  peak VO2 (cardio pulmonary test ; CPX)

SECONDARY OUTCOMES:
remodeling of atrium by the new onset AF in heart failure patients The change of LV function and functional capacity according to the rhythm in patients with HF and new onset AF | 1 years late
  Echo cardiography (LV ejection fraction, LV wall thickness, LV mass index, LA dimension, LA appendage velocity, E/E'), EKG, 24 hours Holter recording
remodeling of ventricle by the new onset AF in heart failure patients The change of LV function and functional capacity according to the rhythm in patients with HF and new onset AF | 1 years late
  Echo cardiography (LV ejection fraction, LV wall thickness, LV mass index, LA dimension, LA appendage velocity, E/E'), EKG, 24 hours Holter recording

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea